CLINICAL TRIAL: NCT06607367
Title: REscuing Bone Marrow Function in Patients with AplaStic AnaEmia and Bone Marrow FaiLure Post AllogEneiC Transplantation 2
Acronym: RESELECT2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.231
Record Dates: First submitted 2024-09-15; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Poor Graft Function; Aplastic Anemia Idiopathic
MeSH Terms: conditions — Anemia, Aplastic | interventions — ruxolitinib; eltrombopag

STUDY DESIGN:
Intervention Model Description: Single group study with historic control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ruxolitinib and Eltrombopag (Experimental): Ruxolitinib at a dose of 10mg BD and Eltrombopag at a dose of 50mg Dose adjustments may be required based on lack of efficacy, or thrombocytopenia may occur as per the study protocol .
  Interventions: Drug: Ruxolitinib (JAKAVI®); Drug: Eltrombopag (Revolade®)

INTERVENTIONS:
Drug: Ruxolitinib (JAKAVI®) — Initial starting dose will be 10mg BD
Drug: Eltrombopag (Revolade®) — Initial starting dose will be 50mg daily

SUMMARY:
Allogeneic stem cell transplantation involves the transplanting of donor blood stem cells into a recipient, this is performed mainly for the treatment of blood cancers. The bone marrow is the organ that produces all blood cells and allogeneic stem cell transplantation results in the replacement of abnormal recipient bone marrow with donor blood cells as well as the production of donor immune cells from the donor bone marrow. The production of donor immune cells will hopefully lead to an immune response directed at any persisting cancerous cells leading to their eradication. As such, one of the key measures of success of a transplant is establishment of donor engraftment.

Engraftment is considered successful when the patient has normal blood cell counts on routine laboratory testing as well as confirmation that the blood cells are being produced by donor bone marrow cells. Confirming donor blood cell production is done by a process called chimerism. Poor graft function (PGF) is a complication of allogeneic stem cell transplantation related to engraftment, manifested by low blood counts despite complete donor chimerism. This has significant consequences for the patient leaving them susceptible to infection because of low white blood cells and bleeding because of low platelets (the cell components that are important for blood clotting). There is currently no established treatment for this condition and patients with this condition who do not recover have a poor survival.

Aplastic anaemia (AA) is a rare autoimmune condition that results in a patient's own immune system attacking important components of their bone marrow resulting in low blood counts. The current treatments for AA include suppressing the immune system or a bone marrow transplant, however long term survival for patients who do not respond to these treatments or relapse is poor and more effective treatments are required.

There is emerging evidence that demonstrates that the components of the immune system are dysfunctional and result in excessive immune activation resulting in suppression of the bone marrow characteristic of PGF. Similar features of immune dysfunction has been demonstrated in AA. Ruxolitinib is a drug that may be able to reduce this excessive immune activation. Eltrombopag is a drug that has been shown to stimulate the production of blood cells. The aim of this study is to evaluate whether the combination of ruxolitinib and eltrombopag is safe and effective in the treatment of PGF and AA.

DETAILED DESCRIPTION:
Study Overview:

This is a, multi-centre, single active arm with historic control arm, phase I/II study that will assess the safety and efficacy of ruxolitinib and eltrombopag in patients with relapse/refractory AA and PGF post alloSCT.

Efficacy will be evaluated using the study endpoints. The study will consist of screening and enrolment (up to 28 days), treatment (12 weeks) and follow up (up to 9 months post enrolment). Therefore, the maximum time on study for a single patient will be a maximum of 12 months.

There will be an initial safety lead in phase of 10 participants. Adverse events will be evaluated by the SMC who will then decide whether the study will proceed to the complete enrolment of 20 participants based on the safety analysis

Treatment:

Upon enrolment, patients in the intervention arm will commence the following treatment: Ruxolitinib at a dose of 10mg BD and Eltrombopag at a dose of 50mg.

Dose adjustments may be required based on lack of efficacy, or thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet ALL of the following:

1. Poor Graft function OR Relapsed/refractory AA

   1. Poor Graft Function defined as follows:≥95% donor chimerism at last reading OR ≥95% CD3 negative chimerism; ≥2 Lineage cytopenias defined as:

      Thrombocytopenia:
      * 30x109 /L from D40-D60 OR
      * 50 x10 9/L from D60 onwards; Neutropenia requiring filgrastim support at any time post D40; Hb less than 80g/L;
   2. Relapsed /Refractory AA defined as: Relapse after stem cell transplant OR relapsed post/refractory to 1st line immunosuppression without an unrelated donor identified.
2. Age ≥18
3. ECOG performance status 0-1
4. Life expectancy greater than 6 months
5. Patient's written informed consent

Exclusion Criteria:

1. Active Grade 3-4 acute GVHD
2. Relapsed or progressive disease on screening bone marrow biopsy or most recent PET imaging.
3. Active second malignancy currently requiring treatment
4. Human Immuno-deficiency Virus (HIV) infection.
5. Any coexisting medical or psychological condition that would preclude participation in the required study procedures.
6. Female patients who are both lactating and breast-feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response at 12 weeks | 12 weeks
  Number of patients with Complete Response (CR) at 12 weeks defined as:
  1. Neutrophils greater than or equal to 1.5x10^9/L
  2. Platelets greater than or equal to 100x10^9/L without use of transfusions or cytokine support
Grade 2 or Higher Non-Haematologic Toxicity | From study enrolment to study completion (maximum of 1 year per subject)
  Rates of grade 2 or higher non haematologic toxicity as graded by the national cancer institute toxicity criteria version 5

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Melbourne Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. Aggregate patient data and final results will be presented in the final report